CLINICAL TRIAL: NCT04849312
Title: Prediction of 30-Day Readmission Using Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Biofourmis Inc. (Industry)
Responsible Party: Principal Investigator, David Levine, Attending Physician, Brigham and Women's Hospital
Other Study IDs: 2017P002583a
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Infection; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulants; Increased
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training: A subset of patients that are used to train the machine learning algorithm.
- Validation: A subset of patients that are "held back" and used to validate the algorithm's accuracy.

SUMMARY:
This is a retrospective observational study drawing on data from the Brigham and Women's Home Hospital database. Sociodemographic and clinic data from a training cohort were used to train a machine learning algorithm to predict the likelihood of 30-day readmission throughout a patient's admission. This algorithm was then validated in a validation cohort.

ELIGIBILITY:
Was a subject in the Brigham and Women's Home Hospital study and has a completed record in the study's database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted at Brigham and Women's Hospital and Brigham and Women's Faulkner Hospital who meet primary diagnosis, age, and residence within 5 mile requirements and are enrolled in home hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
30-Day Readmission [ yes / no ] | From date of admission to 30-days post-discharge (31 to 54 days)
  Unplanned hospital admission within 30 days of having been discharged

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, MD MPH MA, Principal Investigator — Associate Physician
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merrill RK, Ferrandino RM, Hoffman R, Shaffer GW, Ndu A. Machine Learning Accurately Predicts Short-Term Outcomes Following Open Reduction and Internal Fixation of Ankle Fractures. J Foot Ankle Surg. 2019 May;58(3):410-416. doi: 10.1053/j.jfas.2018.09.004. Epub 2019 Feb 23. PMID 30803914
- [Background] Li Q, Yao X, Echevin D. How Good Is Machine Learning in Predicting All-Cause 30-Day Hospital Readmission? Evidence From Administrative Data. Value Health. 2020 Oct;23(10):1307-1315. doi: 10.1016/j.jval.2020.06.009. Epub 2020 Sep 7. PMID 33032774
- [Background] Xue Y, Klabjan D, Luo Y. Predicting ICU readmission using grouped physiological and medication trends. Artif Intell Med. 2019 Apr;95:27-37. doi: 10.1016/j.artmed.2018.08.004. Epub 2018 Sep 10. PMID 30213670
- [Background] Morel D, Yu KC, Liu-Ferrara A, Caceres-Suriel AJ, Kurtz SG, Tabak YP. Predicting hospital readmission in patients with mental or substance use disorders: A machine learning approach. Int J Med Inform. 2020 Jul;139:104136. doi: 10.1016/j.ijmedinf.2020.104136. Epub 2020 Apr 18. PMID 32353752
- [Background] Loreto M, Lisboa T, Moreira VP. Early prediction of ICU readmissions using classification algorithms. Comput Biol Med. 2020 Mar;118:103636. doi: 10.1016/j.compbiomed.2020.103636. Epub 2020 Feb 1. PMID 32174313
- [Background] Bolourani S, Tayebi MA, Diao L, Wang P, Patel V, Manetta F, Lee PC. Using machine learning to predict early readmission following esophagectomy. J Thorac Cardiovasc Surg. 2021 Jun;161(6):1926-1939.e8. doi: 10.1016/j.jtcvs.2020.04.172. Epub 2020 May 29. PMID 32711985
- [Background] Arvind V, London DA, Cirino C, Keswani A, Cagle PJ. Comparison of machine learning techniques to predict unplanned readmission following total shoulder arthroplasty. J Shoulder Elbow Surg. 2021 Feb;30(2):e50-e59. doi: 10.1016/j.jse.2020.05.013. Epub 2020 Jun 9. PMID 32868011